CLINICAL TRIAL: NCT04241172
Title: Rehabilitation of Patients With Total Knee Replacement Through the Immersive Virtual Reality in Aquatic Scenarios
Brief Title: TKR Rehabilitation Through the Immersive Virtual Reality in Aquatic Scenarios
Acronym: HYDROKNEERVANA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to technical issues with the necessary facilities at the participating centers, the PIs have decided to suspend the study until the devices and hydrotherapy pool are fully operational.
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 19/11
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Total Knee Replacement
Keywords: Proprioceptive; Balance; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: patients with total knee prosthesis divided into three groups, to receive a traditional rehabilitation (TR) program, traditional hydrotherapy (TH) or hydrotherapy through immersive virtual reality (HIVR) using Bts-Nirvana
Who Masked: Care Provider
Masking Description: The care providers are not aware about the research study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immersive Virtual Reality (HIVR) (Experimental): The HIVR exercises will be performed using Nirvana system, a medical device based on virtual reality specifically designed to support motor rehabilitation, by projecting aquatic scenarios on the floor that simulates the movement and the noise of the water due to the motor exercise execution by the patient. In particular, the following virtual reality scenarios will be used:
  * "Swimming pool": the environment represents a swimming pool (water and edge). The patient must perform exercises by moving the lower limbs while sitting on a chair. The virtual environment gives the sensation of having the lower limbs immersed in water above the knees;
  * "Water metal": the environment gives the feeling of being immersed in water up to the waist. The subject interacts with the virtual water performing walking exercises and receiving visual and auditory biofeedback.
  Interventions: Device: Experimental: Immersive Virtual Reality (HIVR)
- Traditional Hydrotherapy (TH) (Active Comparator): The TH group exercises will be performed in a swimming pool suitable for hydrotherapy treatments. In particular, patients will perform:
  * exercises with patients sitting on the swimming pool edge with lower limb immersed in the water;
  * flexion-extension of the knee;
  * leg and hip circling;
  * flexion-extension of the ankle;
  * triple flexion;
  * water walking exercises.
  Interventions: Procedure: Traditional Hydrotherapy (TH)
- Traditional Rehabilitation (TR) (Active Comparator): The TR group exercises will be performed in the gym with a physiotherapist. In particular, patients will perform:
  * exercises with a patient sitting on a chair (3 minutes per exercise):
  * flexion-extension of the knee;
  * leg and hip circling;
  * flexion-extension of the ankle;
  * triple flexion;
  * walking (with and without aids).
  Interventions: Procedure: Traditional Rehabilitation (TR)

INTERVENTIONS:
Device: Experimental: Immersive Virtual Reality (HIVR) — the HIVR exercises will be performed using Nirvana system, a medical device based on virtual reality specifically designed to support motor rehabilitation, by projecting aquatic scenarios on the floor that simulates the movement and the noise of the water due to the motor exercise execution by the patient. In particular, the following virtual reality scenarios will be used:
  * "Swimming pool": the environment represents a swimming pool (water and edge). The patient must perform exercises by moving the lower limbs while sitting on a chair. The virtual environment gives the sensation of having the lower limbs immersed in water above the knees;
  * "Water metal": the environment gives the feeling of being immersed in water up to the waist. The subject interacts with the virtual water performing walking exercises and receiving a visual and auditory biofeedback.
  Arms: Immersive Virtual Reality (HIVR)
Procedure: Traditional Hydrotherapy (TH) — The TH group exercises will be performed in a swimming pool suitable for hydrotherapy treatments. In particular, patients will perform:
  * exercises with a patients sitting on the swimming pool edge with lower limb immersed in the water;
  * flexion-extension of the knee;
  * leg and hip circling;
  * flexion-extension of the ankle;
  * triple flexion;
  * water walking exercises.
  Arms: Traditional Hydrotherapy (TH)
Procedure: Traditional Rehabilitation (TR) — The TR group exercises will be performed in the gym with a physiotherapist. In particular, patients will perform:
  * exercises with a patient sitting on a chair (3 minutes per exercise):
  * flexion-extension of the knee;
  * leg and hip circling;
  * flexion-extension of the ankle;
  * triple flexion;
  * walking (with and without aids).
  Arms: Traditional Rehabilitation (TR)

SUMMARY:
This study is a multicenter non-randomized single-blind controlled trial, aimed at investigating the feasibility and efficacy of hydrotherapy based on IVR, for the patients with TKR(Total Knee Replacement), on the function, gait performance, postural balance control, and knee edema reduction. The protocol was draft according to the Consolidated Standards of Reporting Trials (CONSORT ) checklists.

A total of 96patients with total knee prosthesis will be recruited and divided into three groups, to receive a traditional rehabilitation (TR) program, traditional hydrotherapy (TH)or hydrotherapy through immersive virtual reality (HIVR) using Bts-Nirvana. Assessments will be performed at baseline and at the end of treatment.

DETAILED DESCRIPTION:
For the study, inpatients will be taken into consideration. A maximum of 17 treatment sessions will be conducted, divided from 3 to 5 training sessions per week. The treatments will be carried out in groups consisting of 3 patients.

All patients included in the study will perform 45 minutes of traditional rehabilitation treatments, consisted in:

* passive mobilization for the recovery of the complete articular range;
* active work on cycle ergometer;
* muscle strengthening with isometric and isotonic exercises;
* proprioceptive exercises in standing position for load balancing and balance control;
* step training with progressive reduction of walking aids;
* recovery of autonomy in the ascent and descent from the stairs;
* recovery of autonomy in daily life activities. In addition to this common program, specific knee therapy will be performed as provided in the three groups.

Traditional Rehabilitation (TR): the TR group exercises will be performed in the gym with a physiotherapist. In particular, patients will perform:

* exercises with a patient sitting on a chair (3 minutes per exercise):
* flexion-extension of the knee;
* leg and hip circling;
* flexion-extension of the ankle;
* triple flexion;
* walking (with and without aids).

Traditional Hydrotherapy (TH): the TH group exercises will be performed in a swimming pool suitable for hydrotherapy treatments. In particular, patients will perform:

* exercises with patients sitting on the swimming pool edge with lower limb immersed in the water;
* flexion-extension of the knee;
* leg and hip circling;
* flexion-extension of the ankle;
* triple flexion;
* water walking exercises.

Hydrotherapy through Immersive Virtual Reality (HIVR): the HIVR exercises will be performed using Nirvana system, a medical device based on virtual reality specifically designed to support motor rehabilitation, by projecting aquatic scenarios on the floor that simulates the movement and the noise of the water due to the motor exercise execution by the patient. In particular, the following virtual reality scenarios will be used:

* "Swimming pool": the environment represents a swimming pool (water and edge). The patient must perform exercises by moving the lower limbs while sitting on a chair. The virtual environment gives the sensation of having the lower limbs immersed in water above the knees;
* "Water metal": the environment gives the feeling of being immersed in water up to the waist. The subject interacts with the virtual water performing walking exercises and receiving visual and auditory biofeedback.

ELIGIBILITY:
The inclusion criteria are:

* Aged ≤ 85;
* Capacity to consent and to perform the exercises of the specific protocol;
* Patients with total knee prosthesis.

The exclusion criteria are:

* Failure to meet the inclusion criteria;
* Concomitant participation in other studies;
* Unicompartmental knee prostheses;
* Surgery without drainage;
* Wound complications;
* Cognitive disorders;
* Diagnosis of epilepsy;
* Lack of written informed consent;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Time Up & Go Test | At baseline (day 1-T1) and at the end (day 21 -T2) of the treatment.
  Time Up and Go test (TUG): TUG is a test used to determine fall risk and measure the progress of balance, sit to stand and walking. The patient starts in a seated position, then stands up, walks 3 meters, turns around, walks back to the chair and sits down. If a patient took 14 seconds or longer to perform the test he was classified as high-risk for falling

SECONDARY OUTCOMES:
Change in 10-Metre Walking Test (10MWT) | At baseline (day 1-T1) and at the end (day 21 -T2) of the treatment.
  10MWT is used to measure the time (and if required the number of steps) taken for subjects to cover a distance of ten meters from a standing start, when walking at their usual speed, as a measure of the change in aspects of their gait performance

CONTACTS AND LOCATIONS:
Overall Officials: Marco Franceschini, MD, Study Chair — IRCCS San Raffaele; Sanaz Pournajaf, Dr, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffele, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
The protocol for the study will be published shortly.
Supporting Information: Study Protocol
Time Frame: Soon.
Access Criteria: Open Access